CLINICAL TRIAL: NCT04556305
Title: Lifestyle Physical Activity and Cognitive Training Interventions: Preventing Memory Loss in Older Women With Cardiovascular Disease
Brief Title: Lifestyle Physical Activity and Cognitive Training Interventions
Acronym: MindMoves
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 18053104
Record Dates: First submitted 2020-09-04; First posted 2020-09-21 (Actual); Results first posted 2025-03-30 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Cognitive Decline; Cardiovascular Diseases; Cognitive Dysfunction; Cognitive Impairment; Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mind - BrainHQ cognitive training intervention (Experimental): The Mind intervention uses the evidence-based BrainHQ computerized cognitive training program. BrainHQ focuses on improving memory, attention, sensory function, and working memory, and has demonstrated efficacy in improving memory among healthy older adults and adults with heart failure. BrainHQ is tailored to the individual, and program difficulty automatically progresses based on performance. Training occurs during three 30-minute sessions per week, for a total of 36 hours. Participants will complete the BrainHQ program on an iPad tablet, which will be provided to them.
  Interventions: Behavioral: Mind
- Move - lifestyle physical activity intervention (Experimental): The Move intervention is a 24-week evidence-based program based on social cognitive theory. It was originally developed for midlife women and successfully maintained increased physical activity. It has since been tailored for older women with CVD to prevent or delay cognitive decline, and includes: (1) education on the importance of lifestyle physical activity for brain health, (2) increasing lifestyle physical activity while considering CVD, and (3) including a goal for increasing Fitbit "active" minutes (≥ 3 METs or moderate-intensity physical activity) to ensure participants are obtaining the beneficial aerobic fitness effects during periods of lifestyle physical activity. Core elements include a personal lifestyle physical activity goal and five group meetings.
  Interventions: Behavioral: Move
- MindMoves - cognitive training and lifestyle physical activity (Experimental): Participants who are assigned to this condition will complete both the Move lifestyle physical activity program and the Mind BrainHQ cognitive training intervention simultaneously for 24 weeks (see Move and Mind descriptions). Participants will receive both a Fitbit and iPad tablet to complete the combined MindMoves intervention.
  Interventions: Behavioral: Mind; Behavioral: Move
- Usual Care (No Intervention): Participants in the usual care group do not receive any Mind- or Move-related intervention, and will receive their usual care from their cardiology provider.

INTERVENTIONS:
Behavioral: Mind — See arm description.
  Arms: Mind - BrainHQ cognitive training intervention; MindMoves - cognitive training and lifestyle physical activity
Behavioral: Move — See arm description.
  Arms: MindMoves - cognitive training and lifestyle physical activity; Move - lifestyle physical activity intervention

SUMMARY:
Older women with cardiovascular disease (CVD) are at greater risk for memory loss, an important public health issue due to the negative effects to quality of life and health care costs. This research will be the first to examine the independent and combined effects of a lifestyle physical activity intervention and cognitive training on memory performance and memory-related serum biomarkers in this vulnerable population. The investigators will incorporate a practical lifestyle approach that can be delivered in the home and community settings to prevent or delay memory loss in older women with CVD.

DETAILED DESCRIPTION:
Women experience disproportionately high rates of cognitive dysfunction, especially with increasing age, compared to men. Some research suggests that older women have a higher incidence of cognitive dysfunction with greater severity and more rapid decline.Furthermore, cardiovascular disease (CVD) increases the risk for cognitive dysfunction by 29-66% and affects 44 million women in the US.

One particularly distressing type of cognitive dysfunction due to CVD is loss of memory. Memory loss leads to reduced independence, lower quality of life, and higher healthcare costs. To prevent or delay loss of memory among older women with CVD, there is an urgent need to develop lifestyle interventions that can be scaled.

The long-term goal is to create and implement multi-modal lifestyle interventions (interventions that have multiple behavioral components) that will prevent or delay memory loss in older adults. The investigators initially focus on women with CVD due to their high risk. Physical activity interventions and cognitive training each prevent memory loss in healthy older adults.

Thus, the investigators will evaluate the efficacy of MindMoves, a 24-week multi-modal intervention, on memory performance and memory-related serum biomarkers. The investigators will examine the serum biomarkers of brain-derived neurotrophic factor (BDNF), vascular endothelial growth factor (VEGF), and (c) insulin-like growth factor 1 (IGF-1). Data collection will occur at baseline, 24 weeks, 48 weeks, and 72 weeks. MindMoves is a combination of two evidence-based interventions. Mind is the cognitive training program BrainHQ modified to a lifestyle-focused electronic tablet format. Mind improves memory performance in healthy older adults and those with heart failure. Move is a modified lifestyle physical activity intervention from the Women's Lifestyle Physical Activity Program, which the investigators piloted in women with CVD. The investigators recently tested the feasibility of MindMoves.

Using a 2x2 factorial design, the investigators will recruit 254 older women with CVD from cardiology clinics and randomize them to one of the following conditions: (1) Mind, (2) Move, (3) MindMoves, or (4) usual care control. This approach will allow us to evaluate main and interaction effects of Mind and/or Move on memory performance and memory-related biomarkers at 24, 48, and 72 weeks post-baseline.

Specific Aim 1 (primary): Determine the independent and combined efficacies of Mind and Move on memory performance assessed by neurocognitive tests among women ≥ 65 years of age with CVD.

Specific Aim 2 (secondary): Determine the independent and combined efficacies of Mind and Move on memory-related serum biomarkers (BDNF, VEGF, IGF-1) among women ≥ 65 years of age with CVD.

Specific Aim 3 (exploratory): Evaluate depressive symptoms and genetic factors as potential moderators of the association between changes in target behaviors (physical activity and cognitive activity) and health outcomes (memory performance and relevant serum biomarkers).

The investigators hypothesize that Mind and Move individually will each yield benefits to memory. However, it is hypothesized that the combined MindMoves will have a greater impact than the sum of the individual effects. Findings will provide key knowledge about the ability of practical multi-modal lifestyle interventions to target memory in older women with CVD.

ELIGIBILITY:
Inclusion Criteria:

* self-identified as women
* ≥ 65 years old
* read/speak English
* patient in the Rush Heart Center for Women
* history of CVD (e.g., coronary artery disease, hypertension) and receiving guideline-directed medical therapy when appropriate
* no regular moderate-vigorous physical activity (≥ 30 minutes ≥ 3 days per week in the past month)
* no cognitive training program in the past month
* no disabilities preventing regular physical activity (Physical Activity Readiness Questionnaire, which includes cardiac and lung disease symptoms)
* written approval from cardiology provider (Physical Activity Readiness Medical Examination); no self-reported significant hearing loss that interferes with normal conversation
* access to a Bluetooth-capable phone or tablet

Exclusion Criteria:

* symptoms of unstable cardiac or pulmonary disease in the past month (Physical Activity Readiness Questionnaire)
* blood pressure (systolic ≥ 160 or diastolic ≥ 100 mm Hg)
* cognitive status score < 19 on the blind version (for phone administration) of the Montreal Cognitive Assessment (MoCA) consistent with significant cognitive impairment
* diagnosis of a neurological disease found in the electronic health record (e.g., Alzheimer's disease dementia, Parkinson's disease, vascular dementia)
* transient ischemic attack or small-vessel stroke in the past three months
* taking anti-psychotic medication
* diabetes with an A1C ≥ 9.0 within the past six months
* end-stage renal disease on dialysis (Stage 5)

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 253 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2025-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Background] Halloway S, Schoeny ME, Barnes LL, Arvanitakis Z, Pressler SJ, Braun LT, Volgman AS, Gamboa C, Wilbur J. A study protocol for MindMoves: A lifestyle physical activity and cognitive training intervention to prevent cognitive impairment in older women with cardiovascular disease. Contemp Clin Trials. 2021 Feb;101:106254. doi: 10.1016/j.cct.2020.106254. Epub 2020 Dec 29. PMID 33383230
- [Result] Halloway S, Volgman AS, Schoeny ME, Arvanitakis Z, Barnes LL, Pressler SJ, Vispute S, Braun LT, Tafini S, Williams M, Wilbur J. Overcoming Pandemic-Related Challenges in Recruitment and Screening: Strategies and Representation of Older Women With Cardiovascular Disease for a Multidomain Lifestyle Trial to Prevent Cognitive Decline. J Cardiovasc Nurs. 2024 Jul-Aug 01;39(4):359-370. doi: 10.1097/JCN.0000000000001000. Epub 2023 May 11. PMID 37167428
- [Result] Halloway S, Volgman AS, Barnes LL, Schoeny ME, Wilbur J, Pressler SJ, Laddu D, Phillips SA, Vispute S, Hall G, Shakya S, Goodyke M, Auger C, Cagin K, Borgia JA, Arvanitakis ZA. The MindMoves Trial: Cross-Sectional Analyses of Baseline Vascular Risk and Cognition in Older Women with Cardiovascular Disease. J Alzheimers Dis. 2024;100(4):1407-1416. doi: 10.3233/JAD-240100. PMID 39031356
- [Derived] Rogers CA, Yeager C, Schoeny M, Wilbur J, Vispute S, Pressler SJ, Arvanitakis Z, Halloway S. Cognitive Training Intervention Adherence in Older Women with Cardiovascular Disease: A Secondary Analysis of the MindMoves Trial. J Cardiovasc Nurs. 2026 Mar-Apr 01;41(2):E63-E69. doi: 10.1097/JCN.0000000000001291. Epub 2025 Dec 22. PMID 41418039
- [Derived] Halloway S, Schoeny ME, Arvanitakis Z, Volgman AS, Pressler SJ, Vispute S, Wilhelm K, Borgia JA, Wilbur J, Barnes LL. A multidomain trial for cognition in women with cardiovascular disease. Alzheimers Dement. 2025 Jun;21(6):e70285. doi: 10.1002/alz.70285. PMID 40511694

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from two cardiology clinics (one at an academic medical center and one at a nearby community hospital affiliated with the academic medical center) in an urban Midwest area. The study was conducted from 2020 to 2024 in Chicago, Illinois, with enrollment from October 2020 to May 2022 (planned target enrollment achieved), and a final follow-up January 2024.
Pre-assignment Details: A total of 24 cohorts (12 cohorts per each of the two clinic sites) of 10-11 participants each were recruited sequentially prior to baseline assessment. Cluster randomization was used to assign cohorts to cells due to the Move intervention being group-based. Following randomization, the intervention condition was revealed and started at the intervention orientation.
Period: Overall Study
Arm/Group | Mind - BrainHQ Cognitive Training Intervention | Move - Lifestyle Physical Activity Intervention | MindMoves - Cognitive Training and Lifestyle Physical Activity | Usual Care
Started | 64 | 61 | 64 | 64
Completed | 54 | 57 | 54 | 55
Not Completed | 10 | 4 | 10 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mind - BrainHQ Cognitive Training Intervention | Move - Lifestyle Physical Activity Intervention | MindMoves - Cognitive Training and Lifestyle Physical Activity | Usual Care | Total
Number analyzed (Participants) | 64 | 61 | 64 | 64 | 253
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.3 (6.5) | 71.8 (5.7) | 72.5 (5.2) | 72.4 (5.8) | 72.8 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 61 | 64 | 64 | 253
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Latina/Hispanic | 2 | 1 | 3 | 1 | 7
  Asian | 0 | 0 | 1 | 0 | 1
  Non-Hispanic Black or African American | 26 | 26 | 25 | 23 | 100
  Non-Hispanic White | 35 | 34 | 34 | 40 | 143
  Unknown or Not Reported | 1 | 0 | 1 | 0 | 2
Highest education level - College graduate [Count of Participants; unit: Participants] | 44 | 35 | 37 | 35 | 151

OUTCOME MEASURES:

1. Primary Outcome: Change in East Boston Memory Test Scores From Baseline to 24 Weeks, 48 Weeks, and 72 Weeks
Description: The East Boston Memory Test is a performance-based neurocognitive test. Participants are read a brief story with 12 key elements. The participants are asked to recall elements immediately and again after three-minute delay. Each score (immediate and delayed recall) has a scale of 0-12, with a higher score indicating better cognitive performance. The total score is an average of the two subscores for immediate and delayed recall. The total score has a scale of 0-12, with a higher score indicating better cognitive performance.
Time Frame: Baseline, and 24 weeks, 48 weeks, and 72 weeks post-baseline
Population: Intent to treat analysis
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mind - BrainHQ Cognitive Training Intervention | Move - Lifestyle Physical Activity Intervention | MindMoves - Cognitive Training and Lifestyle Physical Activity | Usual Care
Number analyzed (Participants) | 64 | 61 | 64 | 64
score on a scale
  Change from baseline to 24 weeks | 0.03 (0.13) | -0.02 (0.13) | 0.01 (0.13) | 0.05 (0.13)
  Change from baseline to 48 weeks | 0.00 (0.13) | 0.04 (0.13) | 0.28 (0.13) | 0.06 (0.13)
  Change from baseline to 72 weeks | 0.07 (0.13) | 0.15 (0.13) | 0.03 (0.13) | 0.23 (0.13)
Statistical Analysis 1: Comparison: Mind - BrainHQ Cognitive Training Intervention vs Move - Lifestyle Physical Activity Intervention vs MindMoves - Cognitive Training and Lifestyle Physical Activity vs Usual Care; Statistical Test 1: Main effect of Mind (MindMoves + Mind vs. Move + Usual Care) for change over time; Test type: Superiority; p = .409, Mixed Models Analysis
Statistical Analysis 2: Comparison: Mind - BrainHQ Cognitive Training Intervention vs Move - Lifestyle Physical Activity Intervention vs MindMoves - Cognitive Training and Lifestyle Physical Activity vs Usual Care; Statistical Test 2: Main effect of Move (MindMoves + Move vs. Mind + Usual Care) for change over time; Test type: Superiority; p = .456, Mixed Models Analysis
Statistical Analysis 3: Comparison: Mind - BrainHQ Cognitive Training Intervention vs Move - Lifestyle Physical Activity Intervention vs MindMoves - Cognitive Training and Lifestyle Physical Activity vs Usual Care; Statistical Test 3: Interaction effect of Mind x Move (MindMoves + Usual Care vs. Mind + Move) for change over time; Test type: Superiority; p = .692, Mixed Models Analysis

2. Primary Outcome: Change in Category Fluency Test Scores From Baseline to 24 Weeks, 48 Weeks, and 72 Weeks
Description: The Category Fluency Test is a performance-based neurocognitive test. Participants are asked to generate examples for two semantic categories (animals, fruits/vegetables) in separate 60-second trials. There are two separate scores (number of animals generated, number of fruits/vegetables generated). A minimum possible score is 0, with an infinite possible maximum score, with a higher score indicating better cognitive performance.
Time Frame: Baseline, and 24 weeks, 48 weeks, and 72 weeks post-baseline
Population: Intent to treat analysis
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mind - BrainHQ Cognitive Training Intervention | Move - Lifestyle Physical Activity Intervention | MindMoves - Cognitive Training and Lifestyle Physical Activity | Usual Care
Number analyzed (Participants) | 64 | 61 | 64 | 64
score on a scale
  Change from baseline to 24 weeks | -0.08 (0.08) | 0.03 (0.08) | 0.04 (0.08) | 0.18 (0.08)
  Change from baseline to 48 weeks | 0.09 (0.08) | 0.06 (0.08) | 0.08 (0.09) | 0.03 (0.08)
  Change from baseline to 72 weeks | 0.04 (0.08) | 0.09 (0.08) | -0.05 (0.09) | 0.09 (0.08)
Statistical Analysis 1: Comparison: Mind - BrainHQ Cognitive Training Intervention vs Move - Lifestyle Physical Activity Intervention vs MindMoves - Cognitive Training and Lifestyle Physical Activity vs Usual Care; Statistical Test 1: Main effect of Mind (MindMoves + Mind vs. Move + Usual Care) for change over time; Test type: Superiority; p = .179, Mixed Models Analysis
Statistical Analysis 2: Comparison: Mind - BrainHQ Cognitive Training Intervention vs Move - Lifestyle Physical Activity Intervention vs MindMoves - Cognitive Training and Lifestyle Physical Activity vs Usual Care; Statistical Test 2: Main effect of Move (MindMoves + Move vs. Mind + Usual Care) for change over time; Test type: Superiority; p = .910, Mixed Models Analysis
Statistical Analysis 3: Comparison: Mind - BrainHQ Cognitive Training Intervention vs Move - Lifestyle Physical Activity Intervention vs MindMoves - Cognitive Training and Lifestyle Physical Activity vs Usual Care; Statistical Test 3: Interaction effect of Mind x Move (MindMoves + Usual Care vs. Mind + Move) for change over time; Test type: Superiority; p = .159, Mixed Models Analysis

3. Primary Outcome: Change in Digit Span Forwards and Backwards Test Scores From Baseline to 24 Weeks, 48 Weeks, and 72 Weeks
Description: The Digit Span Forwards and Backwards Test is a performance-based neurocognitive test. The examiner says a string of numbers (digit span). For Digit Span Forwards, participant recites digit span, gradually increasing in length. Test stops when participant fails to recite digit span of same length twice. For Digit Span Backwards, participant recites digit span backwards. There are two separate scores (Digit Span Forwards correct responses, Digit Span Backwards correct responses). Digit Span Forwards scores can range from 0-16, with higher scores indicating higher cognitive performance. Digit Span Backwards Scores range from 0-14, with higher scores indicating higher cognitive performance. A total score is a sum of the two scores, with a range of 0-30, with higher scores indicating higher cognitive performance.
Time Frame: Baseline, and 24 weeks, 48 weeks, and 72 weeks post-baseline
Population: Intent to treat analysis
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mind - BrainHQ Cognitive Training Intervention | Move - Lifestyle Physical Activity Intervention | MindMoves - Cognitive Training and Lifestyle Physical Activity | Usual Care
Number analyzed (Participants) | 64 | 61 | 64 | 64
score on a scale
  Change from baseline to 24 weeks | -0.14 (0.09) | -0.04 (0.09) | -0.01 (0.09) | -0.12 (0.09)
  Change from baseline to 48 weeks | 0.02 (0.09) | 0.12 (0.09) | 0.19 (0.10) | -0.16 (0.09)
  Change from baseline to 72 weeks | 0.06 (0.10) | 0.18 (0.09) | -0.08 (0.10) | -0.06 (0.09)
Statistical Analysis 1: Comparison: Mind - BrainHQ Cognitive Training Intervention vs Move - Lifestyle Physical Activity Intervention vs MindMoves - Cognitive Training and Lifestyle Physical Activity vs Usual Care; Statistical Test 1: Main effect of Mind (MindMoves + Mind vs. Move + Usual Care) for change over time; Test type: Superiority; p = .078, Mixed Models Analysis
Statistical Analysis 2: Comparison: Mind - BrainHQ Cognitive Training Intervention vs Move - Lifestyle Physical Activity Intervention vs MindMoves - Cognitive Training and Lifestyle Physical Activity vs Usual Care; Statistical Test 2: Main effect of Move (MindMoves + Move vs. Mind + Usual Care) for change over time; Test type: Superiority; p = .130, Mixed Models Analysis
Statistical Analysis 3: Comparison: Mind - BrainHQ Cognitive Training Intervention vs Move - Lifestyle Physical Activity Intervention vs MindMoves - Cognitive Training and Lifestyle Physical Activity vs Usual Care; Statistical Test 3: Interaction effect of Mind x Move (MindMoves + Usual Care vs. Mind + Move) for change over time; Test type: Superiority; p = .430, Mixed Models Analysis

4. Primary Outcome: Change in Oral Trails A/B Tests Scores From Baseline to 24 Weeks, 48 Weeks, and 72 Weeks
Description: First, participants are asked to count from 1 to 25 (Part A). For Part B, the person is asked to verbally recite alternating numbers and letters until they reach 13 and the letter M. The possible scores is a combined time to completion of both Part A and B summed. Possible minimum score is "discontinued" due to failure to complete the test (a zero score). The maximum score is 300 seconds. A lower score (fewer seconds) indicates higher cognitive performance.
Time Frame: Baseline, and 24 weeks, 48 weeks, and 72 weeks post-baseline
Population: Intent to treat analysis
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Mind - BrainHQ Cognitive Training Intervention | Move - Lifestyle Physical Activity Intervention | MindMoves - Cognitive Training and Lifestyle Physical Activity | Usual Care
Number analyzed (Participants) | 64 | 61 | 64 | 64
seconds
  Change from baseline to 24 weeks | 0.29 (0.12) | 0.12 (0.12) | 0.14 (0.12) | 0.17 (0.12)
  Change from baseline to 48 weeks | 0.40 (0.12) | 0.06 (0.12) | 0.09 (0.12) | 0.22 (0.12)
  Change from baseline to 72 weeks | 0.24 (0.12) | 0.29 (0.12) | 0.28 (0.12) | 0.23 (0.12)
Statistical Analysis 1: Comparison: Mind - BrainHQ Cognitive Training Intervention vs Move - Lifestyle Physical Activity Intervention vs MindMoves - Cognitive Training and Lifestyle Physical Activity vs Usual Care; Statistical Test 1: Main effect of Mind (MindMoves + Mind vs. Move + Usual Care) for change over time; Test type: Superiority; p = .772, Mixed Models Analysis
Statistical Analysis 2: Comparison: Mind - BrainHQ Cognitive Training Intervention vs Move - Lifestyle Physical Activity Intervention vs MindMoves - Cognitive Training and Lifestyle Physical Activity vs Usual Care; Statistical Test 2: Main effect of Move (MindMoves + Move vs. Mind + Usual Care) for change over time; Test type: Superiority; p = .107, Mixed Models Analysis
Statistical Analysis 3: Comparison: Mind - BrainHQ Cognitive Training Intervention vs Move - Lifestyle Physical Activity Intervention vs MindMoves - Cognitive Training and Lifestyle Physical Activity vs Usual Care; Statistical Test 3: Interaction effect of Mind x Move (MindMoves + Usual Care vs. Mind + Move) for change over time; Test type: Superiority; p = .915, Mixed Models Analysis

5. Primary Outcome: Change in Digit Ordering Tests Scores From Baseline to 24 Weeks, 48 Weeks, and 72 Weeks
Description: Participants are asked to memorize and immediately recall in ascending order a series of numbers that gradually increase in length with each trial. Possible scores range from 0-16, with a higher score indicating higher cognitive performance.
Time Frame: Baseline, and 24 weeks, 48 weeks, and 72 weeks post-baseline
Population: intent to treat analysis
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mind - BrainHQ Cognitive Training Intervention | Move - Lifestyle Physical Activity Intervention | MindMoves - Cognitive Training and Lifestyle Physical Activity | Usual Care
Number analyzed (Participants) | 64 | 61 | 64 | 64
score on a scale
  Change from baseline to 24 weeks | -0.14 (0.09) | -0.04 (0.09) | -0.01 (0.09) | -0.12 (0.09)
  Change from baseline to 48 weeks | 0.02 (0.09) | 0.12 (0.09) | 0.19 (0.10) | -0.16 (0.09)
  Change from baseline to 72 weeks | -0.06 (0.10) | 0.18 (0.09) | -0.08 (0.10) | -0.06 (0.09)
Statistical Analysis 1: Comparison: Mind - BrainHQ Cognitive Training Intervention vs Move - Lifestyle Physical Activity Intervention vs MindMoves - Cognitive Training and Lifestyle Physical Activity vs Usual Care; Statistical Test 1: Main effect of Mind (MindMoves + Mind vs. Move + Usual Care) for change over time; Test type: Superiority; p = .078, Mixed Models Analysis
Statistical Analysis 2: Comparison: Mind - BrainHQ Cognitive Training Intervention vs Move - Lifestyle Physical Activity Intervention vs MindMoves - Cognitive Training and Lifestyle Physical Activity vs Usual Care; Statistical Test 2: Main effect of Move (MindMoves + Move vs. Mind + Usual Care) for change over time; Test type: Superiority; p = .130, Mixed Models Analysis
Statistical Analysis 3: Comparison: Mind - BrainHQ Cognitive Training Intervention vs Move - Lifestyle Physical Activity Intervention vs MindMoves - Cognitive Training and Lifestyle Physical Activity vs Usual Care; Statistical Test 3: Interaction effect of Mind x Move (MindMoves + Usual Care vs. Mind + Move) for change over time; Test type: Superiority; p = .430, Mixed Models Analysis

6. Secondary Outcome: Change in Brain-derived Neurotrophic Factor (BDNF) Levels From Baseline to 24 Weeks, 48 Weeks, and 72 Weeks
Description: We will obtain blood samples for BDNF. Pretreatment serum or plasma specimens will be prepared using standard techniques and archived at -80°C in aliquots with no specimen subjected to more than two freeze-thaw cycles. All assays performed in a blinded fashion and according to manufacturer's protocol using a 384-well modified method. Luminex FlexMAP 3D will be used with concentrations calculated based on 7-pt standard curves using a 5-parametric fit algorithm in xPONENT v4.0.3. Following recommendations, serum biomarkers will be obtained in the morning (8am-10am) following an 8-hour fast.
Time Frame: Baseline, and 24 weeks, 48 weeks, and 72 weeks post-baseline
Measure: Mean (Standard Error); unit: log-transformed pg/mL
Arm/Group | Mind - BrainHQ Cognitive Training Intervention | Move - Lifestyle Physical Activity Intervention | MindMoves - Cognitive Training and Lifestyle Physical Activity | Usual Care
Number analyzed (Participants) | 64 | 61 | 64 | 64
log-transformed pg/mL
  Change from baseline to 24 weeks | .01 (.04) | .05 (.04) | .05 (.04) | .05 (.04)
  Change from baseline to 48 weeks | .05 (.04) | .05 (.04) | .06 (.04) | .05 (.04)
  Change from baseline to 72 weeks | .01 (.04) | .05 (.04) | -.01 (.04) | .05 (.04)
Statistical Analysis 1: Comparison: Mind - BrainHQ Cognitive Training Intervention vs Move - Lifestyle Physical Activity Intervention vs MindMoves - Cognitive Training and Lifestyle Physical Activity vs Usual Care; Statistical Test 1: Main effect of Mind (MindMoves + Mind vs. Move + Usual Care) for change over time; Test type: Superiority; p = .487, Mixed Models Analysis
Statistical Analysis 2: Comparison: Mind - BrainHQ Cognitive Training Intervention vs Move - Lifestyle Physical Activity Intervention vs MindMoves - Cognitive Training and Lifestyle Physical Activity vs Usual Care; Statistical Test 2: Main effect of Move (MindMoves + Move vs. Mind + Usual Care) for change over time; Test type: Superiority; p = .827, Mixed Models Analysis
Statistical Analysis 3: Comparison: Mind - BrainHQ Cognitive Training Intervention vs Move - Lifestyle Physical Activity Intervention vs MindMoves - Cognitive Training and Lifestyle Physical Activity vs Usual Care; Statistical Test 3: Interaction effect of Mind x Move (MindMoves + Usual Care vs. Mind + Move) for change over time; Test type: Superiority; p = .908, Mixed Models Analysis

7. Secondary Outcome: Change in Vascular Endothelial Growth Factor A (VEGF) Levels From Baseline to 24 Weeks, 48 Weeks, and 72 Weeks
Description: We will obtain blood samples for VEGF. Pretreatment serum or plasma specimens will be prepared using standard techniques and archived at -80°C in aliquots with no specimen subjected to more than two freeze-thaw cycles. All assays performed in a blinded fashion and according to manufacturer's protocol using a 384-well modified method. Luminex FlexMAP 3D will be used with concentrations calculated based on 7-pt standard curves using a 5-parametric fit algorithm in xPONENT v4.0.3. Following recommendations, serum biomarkers will be obtained in the morning (8am-10am) following an 8-hour fast.
Time Frame: Baseline, and 24 weeks, 48 weeks, and 72 weeks post-baseline
Measure: Mean (Standard Error); unit: log-transformed pg/mL
Arm/Group | Mind - BrainHQ Cognitive Training Intervention | Move - Lifestyle Physical Activity Intervention | MindMoves - Cognitive Training and Lifestyle Physical Activity | Usual Care
Number analyzed (Participants) | 64 | 61 | 64 | 64
log-transformed pg/mL
  Change from baseline to 24 weeks | .02 (.03) | .03 (.03) | -.05 (.03) | .00 (.03)
  Change from baseline to 48 weeks | .06 (.03) | .00 (.03) | .03 (.03) | .03 (.03)
  Change from baseline to 72 weeks | .02 (.03) | -.03 (.03) | .03 (.03) | -.03 (.03)
Statistical Analysis 1: Comparison: Mind - BrainHQ Cognitive Training Intervention vs Move - Lifestyle Physical Activity Intervention vs MindMoves - Cognitive Training and Lifestyle Physical Activity vs Usual Care; Statistical Test 1: Main effect of Mind (MindMoves + Mind vs. Move + Usual Care) for change over time; Test type: Superiority; p = .371, Mixed Models Analysis
Statistical Analysis 2: Comparison: Mind - BrainHQ Cognitive Training Intervention vs Move - Lifestyle Physical Activity Intervention vs MindMoves - Cognitive Training and Lifestyle Physical Activity vs Usual Care; Statistical Test 2: Main effect of Move (MindMoves + Move vs. Mind + Usual Care) for change over time; Test type: Superiority; p = .633, Mixed Models Analysis
Statistical Analysis 3: Comparison: Mind - BrainHQ Cognitive Training Intervention vs Move - Lifestyle Physical Activity Intervention vs MindMoves - Cognitive Training and Lifestyle Physical Activity vs Usual Care; Statistical Test 3: Interaction effect of Mind x Move (MindMoves + Usual Care vs. Mind + Move) for change over time; Test type: Superiority; p = .230, Mixed Models Analysis

8. Secondary Outcome: Change in Insulin-like Growth Factor 1 (IGF-1) From Baseline to 24 Weeks, 48 Weeks, and 72 Weeks
Description: We will obtain blood samples for IGF-1. Pretreatment serum or plasma specimens will be prepared using standard techniques and archived at -80°C in aliquots with no specimen subjected to more than two freeze-thaw cycles. All assays performed in a blinded fashion and according to manufacturer's protocol using a 384-well modified method. Luminex FlexMAP 3D will be used with concentrations calculated based on 7-pt standard curves using a 5-parametric fit algorithm in xPONENT v4.0.3. Following recommendations, serum biomarkers will be obtained in the morning (8am-10am) following an 8-hour fast.
Time Frame: Baseline, and 24 weeks, 48 weeks, and 72 weeks post-baseline
Measure: Mean (Standard Error); unit: square root transformed pg/mL
Arm/Group | Mind - BrainHQ Cognitive Training Intervention | Move - Lifestyle Physical Activity Intervention | MindMoves - Cognitive Training and Lifestyle Physical Activity | Usual Care
Number analyzed (Participants) | 64 | 61 | 64 | 64
square root transformed pg/mL
  Change from baseline to 24 weeks | 3.37 (5.92) | 5.26 (5.65) | 6.59 (5.88) | 8.45 (5.85)
  Change from baseline to 48 weeks | 3.25 (6.05) | 4.24 (5.79) | 6.40 (6.05) | -1.52 (5.89)
  Change from baseline to 72 weeks | 7.55 (5.93) | 4.07 (5.75) | -4.42 (5.97) | 2.71 (5.89)
Statistical Analysis 1: Comparison: Mind - BrainHQ Cognitive Training Intervention vs Move - Lifestyle Physical Activity Intervention vs MindMoves - Cognitive Training and Lifestyle Physical Activity vs Usual Care; Statistical Test 1: Main effect of Mind (MindMoves + Mind vs. Move + Usual Care) for change over time; Test type: Superiority; p = .798, Mixed Models Analysis
Statistical Analysis 2: Comparison: Mind - BrainHQ Cognitive Training Intervention vs Move - Lifestyle Physical Activity Intervention vs MindMoves - Cognitive Training and Lifestyle Physical Activity vs Usual Care; Statistical Test 2: Main effect of Move (MindMoves + Move vs. Mind + Usual Care) for change over time; Test type: Superiority; p = .461, Mixed Models Analysis
Statistical Analysis 3: Comparison: Mind - BrainHQ Cognitive Training Intervention vs Move - Lifestyle Physical Activity Intervention vs MindMoves - Cognitive Training and Lifestyle Physical Activity vs Usual Care; Statistical Test 3: Interaction effect of Mind x Move (MindMoves + Usual Care vs. Mind + Move) for change over time; Test type: Superiority; p = .419, Mixed Models Analysis

9. Secondary Outcome: Change in GT3XE-Plus Triaxial Accelerometer Minutes of Moderate Vigorous Physical Activity From Baseline to 24 Weeks, 48 Weeks, and 72 Weeks
Description: The ActiGraph accelerometer is a motion sensor device that provides a valid assessment of physical activity in adult persons during treadmill Moveing/running and daily activity. The accelerometer records vertical accelerations as "counts." Participants are instructed to wear on the hip for seven consecutive days during waking hours only, except while swimming or bathing. To analyze the accelerometer data, we will use the following physical activity intensity cut points: light 100-1,565 counts/min (< 3 METS [metabolic equivalent of task]); moderate 1,566-6,139 (3.0-6.0 METS); vigorous ≥ 6,140 (≥ 6.1 METS). Findings are reported in mean daily minutes of moderate-vigorous physical activity
Time Frame: Baseline, and 24 weeks, 48 weeks, and 72 weeks post-baseline
Measure: Mean (Standard Error); unit: log-transformed minutes
Arm/Group | Mind - BrainHQ Cognitive Training Intervention | Move - Lifestyle Physical Activity Intervention | MindMoves - Cognitive Training and Lifestyle Physical Activity | Usual Care
Number analyzed (Participants) | 64 | 61 | 64 | 64
log-transformed minutes
  Change from baseline to 24 weeks | -.10 (.10) | .03 (.09) | .06 (.10) | .11 (.10)
  Change from baseline to 48 weeks | -.13 (.10) | -.13 (.09) | -.10 (.10) | -.17 (.09)
  Change from baseline to 72 weeks | -.13 (.10) | -.18 (.09) | -.12 (.10) | .03 (.10)
Statistical Analysis 1: Comparison: Mind - BrainHQ Cognitive Training Intervention vs Move - Lifestyle Physical Activity Intervention vs MindMoves - Cognitive Training and Lifestyle Physical Activity vs Usual Care; Statistical Test 1: Main effect of Mind (MindMoves + Mind vs. Move + Usual Care) for change over time; Test type: Superiority; p = .619, Mixed Models Analysis
Statistical Analysis 2: Comparison: Mind - BrainHQ Cognitive Training Intervention vs Move - Lifestyle Physical Activity Intervention vs MindMoves - Cognitive Training and Lifestyle Physical Activity vs Usual Care; Statistical Test 2: Main effect of Move (MindMoves + Move vs. Mind + Usual Care) for change over time; Test type: Superiority; p = .468, Mixed Models Analysis
Statistical Analysis 3: Comparison: Mind - BrainHQ Cognitive Training Intervention vs Move - Lifestyle Physical Activity Intervention vs MindMoves - Cognitive Training and Lifestyle Physical Activity vs Usual Care; Statistical Test 3: Interaction effect of Mind x Move (MindMoves + Usual Care vs. Mind + Move) for change over time; Test type: Superiority; p = .387, Mixed Models Analysis

10. Secondary Outcome: Change in the Two-minute Step Test of Aerobic Fitness Score From Baseline to 24 Weeks, 48 Weeks, and 72 Weeks
Description: This is a test of aerobic fitness that can be performed in a small space using minimal equipment. Participants step in place to a predesignated height for two minutes. This test is correlated with treadmill tests of aerobic fitness. The score is number of valid steps achieved reaching the predesignated height in two minutes.
Time Frame: Baseline, and 24 weeks, 48 weeks, and 72 weeks post-baseline
Measure: Mean (Standard Error); unit: steps
Arm/Group | Mind - BrainHQ Cognitive Training Intervention | Move - Lifestyle Physical Activity Intervention | MindMoves - Cognitive Training and Lifestyle Physical Activity | Usual Care
Number analyzed (Participants) | 64 | 61 | 64 | 64
steps
  Change from baseline to 24 weeks | -3.52 (2.38) | -2.71 (2.27) | -2.69 (2.34) | -5.10 (2.35)
  Change from baseline to 48 weeks | -3.33 (2.44) | -2.33 (2.31) | -5.64 (2.42) | -9.46 (2.32)
  Change from baseline to 72 weeks | -5.42 (2.42) | -2.15 (2.31) | -7.04 (2.34) | -5.16 (2.33)
Statistical Analysis 1: Comparison: Mind - BrainHQ Cognitive Training Intervention vs Move - Lifestyle Physical Activity Intervention vs MindMoves - Cognitive Training and Lifestyle Physical Activity vs Usual Care; Statistical Test 1: Main effect of Mind (MindMoves + Mind vs. Move + Usual Care) for change over time; Test type: Superiority; p = .380, Mixed Models Analysis
Statistical Analysis 2: Comparison: Mind - BrainHQ Cognitive Training Intervention vs Move - Lifestyle Physical Activity Intervention vs MindMoves - Cognitive Training and Lifestyle Physical Activity vs Usual Care; Statistical Test 2: Main effect of Move (MindMoves + Move vs. Mind + Usual Care) for change over time; Test type: Superiority; p = .759, Mixed Models Analysis
Statistical Analysis 3: Comparison: Mind - BrainHQ Cognitive Training Intervention vs Move - Lifestyle Physical Activity Intervention vs MindMoves - Cognitive Training and Lifestyle Physical Activity vs Usual Care; Statistical Test 3: Interaction effect of Mind x Move (MindMoves + Usual Care vs. Mind + Move) for change over time; Test type: Superiority; p = .219, Mixed Models Analysis

11. Secondary Outcome: Change in Self-reported Physical Activity as Assessed by the Community Healthy Activities Model Program for Seniors (CHAMPS) Survey From Baseline to 24 Weeks, 48 Weeks, and 72 Weeks
Description: The Community Health Activities Model Program for Seniors (CHAMPS) is a 30-item self-report questionnaire that assesses the leisure time, household, and transportation physical activity in past two weeks. Participants are asked how long they participate in 30 different activities and at what frequency. Each activity is assigned intensity. Scores include mean minutes per week of light and moderate-vigorous physical activity for both leisure time and household scales (minimum score of 0 minutes and maximum score of 24 hours, with higher scores indicating more time spent in physical activity).
Time Frame: Baseline, and 24 weeks, 48 weeks, and 72 weeks post-baseline
Measure: Mean (Standard Error); unit: log-transformed hours
Arm/Group | Mind - BrainHQ Cognitive Training Intervention | Move - Lifestyle Physical Activity Intervention | MindMoves - Cognitive Training and Lifestyle Physical Activity | Usual Care
Number analyzed (Participants) | 64 | 61 | 64 | 64
log-transformed hours
  Change from baseline to 24 weeks | .36 (.11) | .32 (.11) | .21 (.11) | .26 (.11)
  Change from baseline to 48 weeks | .40 (.11) | .36 (.11) | .21 (.12) | .28 (.11)
  Change from baseline to 72 weeks | .48 (.12) | .46 (.11) | .45 (.12) | .44 (.11)
Statistical Analysis 1: Comparison: Mind - BrainHQ Cognitive Training Intervention vs Move - Lifestyle Physical Activity Intervention vs MindMoves - Cognitive Training and Lifestyle Physical Activity vs Usual Care; Statistical Test 1: Main effect of Mind (MindMoves + Mind vs. Move + Usual Care) for change over time; Test type: Superiority; p = .995, Mixed Models Analysis
Statistical Analysis 2: Comparison: Mind - BrainHQ Cognitive Training Intervention vs Move - Lifestyle Physical Activity Intervention vs MindMoves - Cognitive Training and Lifestyle Physical Activity; Statistical Test 2: Main effect of Move (MindMoves + Move vs. Mind + Usual Care) for change over time; Test type: Superiority; p = .946, Mixed Models Analysis
Statistical Analysis 3: Comparison: Mind - BrainHQ Cognitive Training Intervention vs Move - Lifestyle Physical Activity Intervention vs MindMoves - Cognitive Training and Lifestyle Physical Activity vs Usual Care; Statistical Test 3: Interaction effect of Mind x Move (MindMoves + Usual Care vs. Mind + Move) for change over time; Test type: Superiority; p = .593, Mixed Models Analysis

12. Secondary Outcome: Change in Self-reported Cognitive Activity From Baseline to 24 Weeks, 48 Weeks, and 72 Weeks
Description: Self-report cognitive activity is a self-report questionnaire of participation in nine activities that involve information processing with minimal physical or social demands. Participants rate on a five-point scale. The score is an average of nine items (minimum score of 9, maximum score of 54 with higher scores indicating higher self-reported levels of cognitive activity).
Time Frame: Baseline, and 24 weeks, 48 weeks, and 72 weeks post-baseline
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mind - BrainHQ Cognitive Training Intervention | Move - Lifestyle Physical Activity Intervention | MindMoves - Cognitive Training and Lifestyle Physical Activity | Usual Care
Number analyzed (Participants) | 64 | 61 | 64 | 64
score on a scale
  Change from baseline to 24 weeks | .03 (.07) | .15 (.07) | .08 (.07) | .02 (.07)
  Change from baseline to 48 weeks | .01 (.07) | .21 (.07) | -.04 (.07) | .03 (.07)
  Change from baseline to 72 weeks | -.10 (.07) | .21 (.07) | .12 (.07) | .13 (.07)
Statistical Analysis 1: Comparison: Mind - BrainHQ Cognitive Training Intervention vs Move - Lifestyle Physical Activity Intervention vs MindMoves - Cognitive Training and Lifestyle Physical Activity vs Usual Care; Statistical Test 1: Main effect of Mind (MindMoves + Mind vs. Move + Usual Care) for change over time; Test type: Superiority; p = .092, Mixed Models Analysis
Statistical Analysis 2: Comparison: Mind - BrainHQ Cognitive Training Intervention vs Move - Lifestyle Physical Activity Intervention vs MindMoves - Cognitive Training and Lifestyle Physical Activity vs Usual Care; Statistical Test 2: Main effect of Move (MindMoves + Move vs. Mind + Usual Care) for change over time; Test type: Superiority; p = .245, Mixed Models Analysis
Statistical Analysis 3: Comparison: Mind - BrainHQ Cognitive Training Intervention vs Move - Lifestyle Physical Activity Intervention vs MindMoves - Cognitive Training and Lifestyle Physical Activity vs Usual Care; Statistical Test 3: Interaction effect of Mind x Move (MindMoves + Usual Care vs. Mind + Move) for change over time; Test type: Superiority; p = .107, Mixed Models Analysis

13. Secondary Outcome: Change in GT3XE-Plus Triaxial Accelerometer Minutes of Light Physical Activity From Baseline to 24 Weeks, 48 Weeks, and 72 Weeks
Description: The ActiGraph accelerometer is a motion sensor device that provides a valid assessment of physical activity in adult persons during treadmill Moveing/running and daily activity. The accelerometer records vertical accelerations as "counts." Participants are instructed to wear on the hip for seven consecutive days during waking hours only, except while swimming or bathing. To analyze the accelerometer data, we will use the following physical activity intensity cut points: light 100-1,565 counts/min (< 3 METS [metabolic equivalent of task]); moderate 1,566-6,139 (3.0-6.0 METS); vigorous ≥ 6,140 (≥ 6.1 METS). Findings are reported in mean daily minutes of light physical activity
Time Frame: Baseline, and 24 weeks, 48 weeks, and 72 weeks post-baseline
Measure: Mean (Standard Error); unit: daily minutes
Arm/Group | Mind - BrainHQ Cognitive Training Intervention | Move - Lifestyle Physical Activity Intervention | MindMoves - Cognitive Training and Lifestyle Physical Activity | Usual Care
Number analyzed (Participants) | 64 | 61 | 64 | 64
daily minutes
  Change from baseline to 24 weeks | -10.04 (6.96) | 2.83 (6.76) | 2.13 (7.13) | .09 (6.99)
  Change from baseline to 48 weeks | 6.62 (7.32) | -12.49 (6.80) | -3.84 (7.49) | -3.47 (6.85)
  Change from baseline to 72 weeks | 2.46 (7.18) | -6.40 (6.76) | -8.08 (7.22) | -3.21 (7.13)
Statistical Analysis 1: Comparison: Mind - BrainHQ Cognitive Training Intervention vs Move - Lifestyle Physical Activity Intervention vs MindMoves - Cognitive Training and Lifestyle Physical Activity vs Usual Care; Statistical Test 1: Main effect of Mind (MindMoves + Mind vs. Move + Usual Care) for change over time; Test type: Superiority; p = .244, Mixed Models Analysis
Statistical Analysis 2: Comparison: Mind - BrainHQ Cognitive Training Intervention vs Move - Lifestyle Physical Activity Intervention vs MindMoves - Cognitive Training and Lifestyle Physical Activity vs Usual Care; Statistical Test 2: Main effect of Move (MindMoves + Move vs. Mind + Usual Care) for change over time; Test type: Superiority; p = .085, Mixed Models Analysis
Statistical Analysis 3: Comparison: Mind - BrainHQ Cognitive Training Intervention vs Move - Lifestyle Physical Activity Intervention vs MindMoves - Cognitive Training and Lifestyle Physical Activity vs Usual Care; Statistical Test 3: Interaction effect of Mind x Move (MindMoves + Usual Care vs. Mind + Move) for change over time; Test type: Superiority; p = .710, Mixed Models Analysis

14. Other Pre Specified Outcome: Level and Change in Center for Epidemiologic Studies-Depression Scale Score From Baseline to 24 Weeks, 48 Weeks, and 72 Weeks.
Description: Depressive symptoms will be evaluated as a potential moderator. The Center for Epidemiologic Studies-Depression Scale (20 items scored 0-3) assesses symptoms of depressed mood, feelings of guilt and worthlessness, feelings of helplessness and hopelessness, psychomotor retardation, loss of appetite, and sleep disturbance. Participants who score ≥ 16 will be referred to their primary/ psychiatric provider for further evaluation and treatment. Scores range from 0-60, with higher score indicating more depressive symptoms.
Time Frame: Baseline, and 24 weeks, 48 weeks, and 72 weeks post-baseline
Measure: Mean (Standard Error); unit: log-transformed score on a scale
Arm/Group | Mind - BrainHQ Cognitive Training Intervention | Move - Lifestyle Physical Activity Intervention | MindMoves - Cognitive Training and Lifestyle Physical Activity | Usual Care
Number analyzed (Participants) | 64 | 61 | 64 | 64
log-transformed score on a scale
  Change from baseline to 24 weeks | -.07 (.11) | .09 (.11) | .00 (.11) | .16 (.11)
  Change from baseline to 48 weeks | -.18 (.11) | -.07 (.11) | -.05 (.11) | .07 (.11)
  Change from baseline to 72 weeks | .02 (.11) | -.08 (.11) | -.24 (.11) | .00 (.11)
Statistical Analysis 1: Comparison: Mind - BrainHQ Cognitive Training Intervention vs Move - Lifestyle Physical Activity Intervention vs MindMoves - Cognitive Training and Lifestyle Physical Activity vs Usual Care; Statistical Test 1: Main effect of Mind (MindMoves + Mind vs. Move + Usual Care) for change over time; Test type: Superiority; p = .491, Mixed Models Analysis
Statistical Analysis 2: Comparison: Mind - BrainHQ Cognitive Training Intervention vs Move - Lifestyle Physical Activity Intervention vs MindMoves - Cognitive Training and Lifestyle Physical Activity vs Usual Care; Statistical Test 2: Main effect of Move (MindMoves + Move vs. Mind + Usual Care) for change over time; Test type: Superiority; p = .444, Mixed Models Analysis
Statistical Analysis 3: Comparison: Mind - BrainHQ Cognitive Training Intervention vs Move - Lifestyle Physical Activity Intervention vs MindMoves - Cognitive Training and Lifestyle Physical Activity vs Usual Care; Statistical Test 3: Interaction effect of Mind x Move (MindMoves + Usual Care vs. Mind + Move) for change over time; Test type: Superiority; p = .279, Mixed Models Analysis

15. Other Pre Specified Outcome: Apolipoprotein [APOE]- ε4 Allele
Description: Potential moderator. Candidate gene analysis with DNA extraction from whole blood samples using an Autogen DNA isolation kit (Qiagen, Venlo, Netherlands). Participants will be characterized by APOE genotype and subdivided into two groups of patients in whom the APOE ε4 allele was absent or present.
Time Frame: Baseline
Population: The number of participants analyzed represents the total of number of participants for whom blood was drawn and successfully analyzed to determine APOE genotype.
Measure: Count of Participants; unit: Participants
Arm/Group | Mind - BrainHQ Cognitive Training Intervention | Move - Lifestyle Physical Activity Intervention | MindMoves - Cognitive Training and Lifestyle Physical Activity | Usual Care
Number analyzed (Participants) | 60 | 60 | 63 | 63
Participants
  Count of participants with APOE ε4 allele present | 10 | 16 | 18 | 18
  Count of participants with APOE ε4 allele absent | 50 | 44 | 45 | 45

16. Other Pre Specified Outcome: Brain-derived Neurotrophic Factor (BDNF) Val66Met Polymorphism
Description: Potential moderator. Val66Met polymorphism in the BDNF gene assessed using candidate genotyping. The BDNF gene locus is located on Chromosome 11. BDNF Met positive genotypes are heterozygous Val/Met or homozygous Met/Met. Results will be reported as presence of Met allele or absence of Met allele
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Mind - BrainHQ Cognitive Training Intervention | Move - Lifestyle Physical Activity Intervention | MindMoves - Cognitive Training and Lifestyle Physical Activity | Usual Care
Number analyzed (Participants) | 64 | 61 | 64 | 64
Participants
  Met allele present | 17 | 9 | 18 | 9
  Met allele absent | 47 | 52 | 46 | 55

ADVERSE EVENTS:
Time Frame: From baseline through follow-up data collection at 72 weeks
Arm/Group | Mind - BrainHQ Cognitive Training Intervention | Move - Lifestyle Physical Activity Intervention | MindMoves - Cognitive Training and Lifestyle Physical Activity | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/64 | 2/61 | 1/64 | 1/64
Serious Adverse Events (participants affected / at risk) | 1/64 | 1/61 | 0/64 | 2/64
Other Adverse Events (participants affected / at risk) | 4/64 | 6/61 | 6/64 | 5/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mind - BrainHQ Cognitive Training Intervention (N=64) | Move - Lifestyle Physical Activity Intervention (N=61) | MindMoves - Cognitive Training and Lifestyle Physical Activity (N=64) | Usual Care (N=64)
Hospitalization (General disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mind - BrainHQ Cognitive Training Intervention (N=64) | Move - Lifestyle Physical Activity Intervention (N=61) | MindMoves - Cognitive Training and Lifestyle Physical Activity (N=64) | Usual Care (N=64)
Elevated depressive symptoms (Psychiatric disorders) | 2 (2) | 3 (3) | 3 (3) | 4 (4) — Participants who score 16 or higher on the CES-D at any time point. Pt was referred to their primary or psychiatric provider for further evaluation and treatment.
Chest pain (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Patients who experience angina or chest pain with physical activity or data collection
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 3 (3) | 1 (1) — Participants may experience joint pain (e.g., knee or hip joint pain) when increasing physical activity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-01-26): https://cdn.clinicaltrials.gov/large-docs/05/NCT04556305/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-26): https://cdn.clinicaltrials.gov/large-docs/05/NCT04556305/SAP_001.pdf
  • Informed Consent Form (2021-01-26): https://cdn.clinicaltrials.gov/large-docs/05/NCT04556305/ICF_002.pdf